CLINICAL TRIAL: NCT01075100
Title: Phase II Trial of Ixabepilone Plus Carboplatin in Patients With Metastatic Breast Cancer: The ECLIPSE Study
Brief Title: Ixabepilone + Carboplatin Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08007
Record Dates: First submitted 2010-01-14; First posted 2010-02-24 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic; breast; cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — ixabepilone; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weekly Ixabepilone +carboplatin (Experimental): Subjects will receive ixabepilone and carboplatin on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: Ixabepilone; Drug: Carboplatin

INTERVENTIONS:
Drug: Ixabepilone — 20 mg/m2 on Days 1 and 8
  Other Names: Ixempra; azaepothilone B
Drug: Carboplatin — carboplatin AUC=2.5 on Days 1 and 8
  Other Names: Paraplatin

SUMMARY:
Ixabepilone adds significantly to the antitumor effectiveness of capecitabine in both ER+ and triple negative breast cancer. Ixabepilone has substantial antitumor activity in taxane-refractory patients and novel combinations are needed in this poor prognosis population. Carboplatin in combination with gemcitabine or paclitaxel has activity in metastatic breast cancer (MBC); there is also demonstrated activity of the gemcitabine/carboplatin combination in the ER+ versus triple negative subsets. A Phase I study of ixabepilone plus carboplatin in solid tumor patients demonstrated the safety of this combination at the doses and schedule proposed for this Phase II trial (BMS data on file).

DETAILED DESCRIPTION:
This is a Phase II, open label, nonrandomized, parallel, noncomparative, study of 2 groups (as stratified below). All patients will receive ixabepilone 20 mg/m2 on Days 1 and 8 and carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle. Patients will be stratified by either hormone receptor positive [ER+/PR+/HER2-, ER+/PR-/HER2-, ER-/PR+/HER2-]- (n=50) or triples negative ER-/PR-/HER2- (n=53). If one group fulfills their accrual goal first, registration into that strata will be stopped and only patients meeting stratification requirements for the other group will be registered.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients will be eligible for inclusion in this study if they meet all of the following criteria:

1. Has measurable metastatic and or locally unresectable breast cancer with documented HER2 negative (-) disease
2. Has at least 1 measurable lesion per RECIST criteria (lesions that can be accurately measured in at least 1 dimension (longest diameter (LD) to be recorded) as ≥20 mm with conventional techniques (CT, MRI, X-ray) or as ≥10 mm with spiral CT scan). Irradiated lesions cannot be used to assess response but can be used to assess progression.
3. Has received up to 2 (0 to 2) prior chemotherapy regimens for metastatic disease with the following conditions:

   •Has had no prior treatment with ixabepilone or platinum agents
4. Has had no adjuvant chemotherapy within the 6 months prior to study, but may have received prior anthracyclines and/or taxanes as adjuvant chemotherapy
5. 3 weeks or more have elapsed since last chemotherapy treatment and any related toxicities have resolved to <Grade 1; at least 30 days must have passed since any investigational product has been administered and associated toxicities must have resolved to <Grade 1 (if applicable).
6. Has an ECOG Performance Status (PS) 0-2
7. Is ≥18 years of age
8. Has a life expectancy of at least 12 weeks
9. Has laboratory values of:

   White blood cell (WBC) count ≥3000 x 106/L Absolute neutrophil count (ANC) ≥1500 x 106/L Hemoglobin ≥9 g/dL Total bilirubin ≤1x upper limit of normal (ULN) AST and ALT ≤2.5 x ULN Alkaline phosphatase ≤2.5 x ULN; up to 5xULN if elevation is due to bone disease Serum creatinine ≤1.5 mg/dL Calculated creatinine clearance >50 mL/min (based on Cockroft and Gault method [Appendix III]) Platelet count ≥100,000 x 106/L
10. If patient has had radiation therapy, it has been completed >3 weeks prior to the start of study treatment. NOTE: Previously irradiated lesions will not be evaluable. However, these patients will still be eligible.
11. Has a negative serum pregnancy test within 7 calendar days prior to registration (female patients of childbearing potential [not surgically sterilized and between menarche and 1 year postmenopause
12. If fertile, patient (male or female) has agreed to use an acceptable method of birth control to avoid pregnancy for the duration of the study and for a period of 3 months thereafter
13. Has signed the most recent Patient Informed Consent Form
14. Has signed a Patient Authorization Form Note: Having tissue available is not an inclusion criterion in this study; however, available tissue will be collected (see Section 8) if possible.

Exclusion Criteria:

A patient will be excluded from this study if he or she meets any of the following criteria:

1. Had prior treatment with ixabepilone or other epothilones
2. Had prior radiation to ≥30% of major bone marrow containing areas (pelvis, lumbar spine)
3. Has ER+ and/or PR+ disease that has not progressed on hormone therapy, unless the patient has life-threatening or rapidly progressing visceral disease
4. Has HER2+ disease (IHC staining of 3+ [uniform, intense membrane staining of >30% of invasive tumor cells]), a FISH result of more than 6 HER2 gene copies per nucleus or a FISH ratio (HER2 gene signals to chromosome 17 signals of >2.2)
5. Has only lytic bone disease or nonmeasurable disease only
6. Has a known, prior, severe (NCI CTCAE Grade 3-4) history of hypersensitivity reaction to a drug formulated in Cremophor®EL (polyoxyethylated castor oil) or has history of severe allergic reactions to cisplatin or other platinum-containing compounds
7. Has been treated previously with a platinum-containing agent
8. Is receiving concurrent immunotherapy, hormonal therapy, or radiation therapy. Washout periods for these prior therapies are specified in Section 5.
9. Is receiving concurrent investigational therapy or has received such therapy within the 30 days prior to dosing Day 1
10. Has neuropathy (motor or sensory) >Grade 1
11. Has evidence of CNS involvement requiring radiation or steroid treatment. Patients with stable brain metastases who are off steroids at least 2 weeks are eligible.
12. Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
13. Has clinically relevant coagulopathy either secondary to hepatic dysfunction or an underlying condition requiring therapeutic anticoagulation (specifically, A-fib, history of DVT). A daily aspirin or Plavix for CAD are permitted.
14. Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs
15. Is a pregnant or breast feeding woman
16. Is unable to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Osborne, MD, Principal Investigator — US Oncology
Locations (59):
- United States (59):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Southwest Cancer care, Murrieta, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Institute - New Hope, Hudson, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Florida Institute of Research, Medicine & Surgery, Ocoee, Florida
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Carmel, Indiana
  - Alliance Hematology Oncology, P.A., Westminster, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Maryland Oncology Hematology, PA The Medical Pavillion at Howard County, Columbia, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Cancer Center, LLC, Kansas City, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Comprehensive Cancer Care Centers of Nevada, Henderson, Nevada
  - Hematology-Oncology Associates of Northern NJ, PA Carol G. Simon Cancer Center, Morristown, New Jersey
  - Ruth Oratz MD, New York, New York
  - Interlakes Oncology & Hematology, P.C, Rochester, New York
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Dayton Oncology & Hematology, P.A. Greater Dayton Cancer Center, Kettering, Ohio
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology - Abilene, Abilene, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology Medical City Dallas, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology- Denton South, Denton, Texas
  - Texas Oncology-Fort Worth 12 Ave, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology- Lewisville, Lewisville, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology-McAllen South Second Street, McAllen, Texas
  - Texas Oncology-Mesquite, Mesquite, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology- Odessa West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Cancer Care Centers of South Texas-HOAST, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology-Waco, Waco, Texas
  - Texas Oncology Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Columbia Basin Hematology & Oncology, Kennewick, Washington
  - Puget Sound Cancer Centers, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Evergreen Hematology & Oncology, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Raleigh Regional Cancer Center dba Beckley Oncology Associates Inc., Beckley, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Triple Negative: ER-/PR-/HER2- patients who received Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
- HR Positive: ER+/PR+/HER2-, or ER+/PR-/HER2-, or ER-/PR+/HER2- patients who received receive Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
Period: Overall Study
Arm/Group | Triple Negative | HR Positive
Started | 49 | 54
Completed | 0 | 1
Not Completed | 49 | 53
Not completed — Adverse Event | 15 | 18
Not completed — Patient Request | 4 | 4
Not completed — Investigator Request | 2 | 1
Not completed — Disease Progression | 25 | 29
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Triple Negative: ER-/PR-/HER2- patients who received receive Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Triple Negative | HR Positive | Total
Number analyzed (Participants) | 49 | 54 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.0) | 56.7 (10.6) | 55.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 33 | 39 | 72
  Hispanic | 2 | 2 | 4
  Hawaiian | 0 | 1 | 1
  Black | 14 | 10 | 24
  Asian | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 54 | 103

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Evaluate the objective response rate calculated as CR+ PR in the population evaluable for response, as well as the 2 subgroups (hormone receptor positive [ER+/PR+/HER2-, ER+/PR-/HER2-, ER-/PR+/HER2-]) and ER-/PR-HER2-, separately).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 months
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HR Positive: ER+/PR+/HER2-, or ER+/PR-/HER2-, or ER-/PR+/HER2- patients who received Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 46 | 53
percentage of participants | 30.4 [17.7 to 45.8] | 34 [21.5 to 48.3]

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) defined as objective response rate (ORR, CR + PR) + SD >= 6 months
Time Frame: 24 months
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 46 | 53
percentage of participants | 41.3 [27.0 to 56.8] | 56.6 [42.3 to 70.2]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 24 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 49 | 54
months | 7.6 [4.3 to 8.4] | 7.6 [4.2 to 9.8]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 24 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- HR Positive: ER+/PR+/HER2-, or ER+/PR-/HER2-, or ER-/PR+/HER2- patients who receive Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 49 | 54
months | 12.5 [10.2 to 14.2] | 17.9 [14.4 to 22.4]

5. Secondary Outcome: Time to Response
Description: For patients who achieve a major objective response (CR or PR) the time to response will be assessed as the date of registration to the date of response.
Time Frame: 24 months
Population: Patients who achieve a major objective response (CR or PR).
Measure: Median (Full Range); unit: months
Groups:
- Triple Negative: ER-/PR-/HER2- patients who receive Ixabepilone 20 mg/m2 on Days 1 and 8 and Carboplatin AUC=2.5 on Days 1 and 8 of each 21-day cycle.
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 14 | 18
months | 1.27 [0.92 to 3.98] | 1.60 [1.12 to 8.95]

6. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are first met for CR/PR until the first date that recurrent or progressive disease is objectively documented.
Time Frame: 30 months
Population: Patients who achieved CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Triple Negative | HR Positive
Number analyzed (Participants) | 14 | 18
months | 6.68 [2.43 to 20.4] | 5.92 [1.84 to 25.6]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Triple Negative | HR Positive
Serious Adverse Events (participants affected / at risk) | 10/48 | 5/53
Other Adverse Events (participants affected / at risk) | 44/48 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple Negative (N=48) | HR Positive (N=53)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
APPETITE DECREASED (Gastrointestinal disorders) | 0 (0) | 1 (1)
BACTERIAL RESISTANCE (Infections and infestations) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 4 (4) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 4 (4) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
EMBOLISM PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEVER (General disorders) | 1 (1) | 1 (1)
FIBRILLATION ATRIAL (Cardiac disorders) | 1 (1) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOTENSION (Cardiac disorders) | 1 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATION RATE DECREASED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RIGORS (General disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
VOLUME BLOOD DECREASED (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1)
WEAKNESS GENERALIZED (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple Negative (N=48) | HR Positive (N=53)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6) | 5 (6)
ALLERGIC REACTION (Immune system disorders) | 3 (3) | 5 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (16) | 20 (22)
ANEMIA (Blood and lymphatic system disorders) | 27 (58) | 28 (103)
ANOREXIA (Gastrointestinal disorders) | 6 (8) | 13 (18)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6)
CHILLS (General disorders) | 3 (3) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 13 (17)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 7 (12)
DIARRHEA (Gastrointestinal disorders) | 13 (18) | 15 (22)
DIZZINESS (Nervous system disorders) | 2 (2) | 4 (4)
DYSGUESIA (Gastrointestinal disorders) | 6 (6) | 8 (12)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
EDEMA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 18 (29) | 31 (58)
FEVER (General disorders) | 3 (3) | 3 (3)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 2 (2) | 3 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
LEUCOPENIA (Blood and lymphatic system disorders) | 6 (13) | 14 (58)
MUCOSITIS (Infections and infestations) | 1 (1) | 3 (4)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (8) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (7)
NAUSEA (Gastrointestinal disorders) | 23 (40) | 31 (47)
NEUROPATHY (Nervous system disorders) | 22 (35) | 27 (51)
NEUTROPENIA (Blood and lymphatic system disorders) | 31 (99) | 39 (184)
PAIN (General disorders) | 2 (2) | 5 (6)
PAIN BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 (44) | 25 (65)
VOMITING (Gastrointestinal disorders) | 8 (12) | 19 (26)
WEAKNESS (General disorders) | 4 (6) | 2 (2)
WEIGHT LOSS (General disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No